CLINICAL TRIAL: NCT01627444
Title: Ear Acupuncture for Anxiety in Mothers of Very Low Birth Weight Infants
Brief Title: Acupuncture in Mothers of Very Low Birth Weight Infants
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mariana Haddad, Doctorate Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Acupuncture_doctorate
Record Dates: First submitted 2012-06-20; First posted 2012-06-25 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Anxiety
Keywords: Acupuncture; Anxiety; Human Milk; Very low birth weight infants; Mother of very low birth weight infants
MeSH Terms: conditions — Anxiety Disorders | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- ear acupuncture (Experimental)
  Interventions: Procedure: Ear acupuncture
- Placebo acupuncture (Placebo Comparator): No needle insertion, only stickers on acupuncture points.
  Interventions: Procedure: Ear acupuncture

INTERVENTIONS:
Procedure: Ear acupuncture — Ear acupuncture based on Chinese Map: ShenMen, Anxiety 1 and 2, Tension, Muscular relaxation.

SUMMARY:
Does ear acupuncture reduce anxiety in mother of very low birth weight infants?

ELIGIBILITY:
Inclusion Criteria:

* can read and write in portuguese

Exclusion Criteria:

* breastfeeding contraindication
* use of lactogogues

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Reduced anxiety | at least 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário de Londrina, Londrina, Paraná, Brazil